CLINICAL TRIAL: NCT04619914
Title: Comparison of the Effect of Clomiphene Citrate Plus Estradiol Valerate Versus Letrozole on Endometrial Thickness and Pregnancy Rate in Infertile Women With Polycystic Ovarian Syndrome
Brief Title: the Effect of Clomiphene Citrate Plus Estradiol Valerate Versus Letrozole on Endometrial Thickness and Pregnancy Rate in Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laylay Mohammed Khalleefah Alhibshi (Other Government)
Responsible Party: Sponsor-Investigator, Laylay Mohammed Khalleefah Alhibshi, M.B.B.CH , Faculty of Medicine, Aljabal -Algharbi university - Libya, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB# 5057/19-12-2018
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Endometrial Thickness; Pregnancy Rate
Keywords: Letrozole; clomiphene Citrate; PCOS; Endometrial thickness
MeSH Terms: interventions — Clomiphene; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (clomiphene citrate & estradiol group) (Experimental): included 35 anovulatory PCO patients who received clomiphene citrate (Clomid; Aventis pharma S.AE, Global Napi pharmaceuticals, Cairo, Egypt) 100 mg daily from cycle day 3 to 7 with estradiol valerate 4-mg (two white tablets of cyclopregynova) from cycle day 8 to 14
  Interventions: Drug: Clomid; Aventis pharma S.AE, Global Napi pharmaceuticals, Cairo, Egypt
- Group B (Letrozole group) (Experimental): included 35 anovulatory PCO patients who received letrozole (Femara; Novartis pharma AG, Basle, Switzerland) 5 mg daily from cycle day 3 to day 7.
  Interventions: Drug: letrozole (Femara; Novartis pharma AG, Basle, Switzerland)

INTERVENTIONS:
Drug: Clomid; Aventis pharma S.AE, Global Napi pharmaceuticals, Cairo, Egypt — CLOMID (clomiphene citrate tablets USP) is an orally administered, nonsteroidal, ovulatory stimulant designated chemically as 2-[p-(2-chloro-1,2-diphenylvinyl)phenoxy] triethylamine citrate (1:1)
  Arms: Group A (clomiphene citrate & estradiol group)
Drug: letrozole (Femara; Novartis pharma AG, Basle, Switzerland) — Letrozole, or CGS 20267, is an oral non-steroidal type II aromatase inhibitor. It is a third generation aromatase inhibitor like exemestane and anastrozole, meaning it does not significantly affect cortisol, aldosterone, and thyroxine.
  Arms: Group B (Letrozole group)

SUMMARY:
The present randomized double blind study has been carried out in Gynecology and Obstetrics Department, Faculty of Medicine, Zagazig university on 70 women were previously received clomiphene citrate alone as management of infertile anovulatory PCOS women, but giving improper endometrial thickness < 7mm during the period from March 2019 to September 2019

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome (PCOS) is the most common endocrine disorder in infertile women. Infertility affects 40% of women with PCOS. Understanding the main causes of infertility and selecting an appropriate treatment plan is a diagnostic and therapeutic priority The aim of this work was to compare the effect of Clomiphene citrate plus Estradiol Valerate versus Letrozole on endometrial thickness and pregnancy rate in infertile PCOS women underwent ovulation induction

The study was designed as a randomized double blind study using a computer-generated randomization list and sequentially numbered opaque sealed envelopes, each containing the allocation information written on a card. Envelopes were opened sequentially by a study nurse to allocate patients to the assigned group. These patients were divided into two groups:

1. Group A (clomiphene citrate & estradiol group): included 35 anovulatory PCO patients who received clomiphene citrate (Clomid; Aventis pharma S.AE, Global Napi pharmaceuticals, Cairo, Egypt) 100 mg daily from cycle day 3 to 7 with estradiol valerate 4-mg (two white tablets of cyclopregynova) from cycle day 8 to 14.
2. Group B (Letrozole group): included 35 anovulatory PCO patients who received letrozole (Femara; Novartis pharma AG, Basle, Switzerland) 5 mg daily from cycle day 3 to day 7.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-35 years old with complete infertility workup
* patients diagnosed as having PCOs women
* Normal semen analysis

Exclusion Criteria:

* Patients with male factor infertility, hyperprolactinemia, thyroid disorder.
* Patients with any tubal pathology or uterine pathology.
* Contraindication of ovulation induction, (Multiple ovarian cysts or allergy to inducing agent "clomid").
* Known or suspected pelvic infection (PID).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
the endometrial thickness | up to 24 weeks
  Thickness was measured by placing electronic calipers on the outer walls of the endometrium at its widest diameter as seen in the longitudinal axis of the uterine body

SECONDARY OUTCOMES:
the ovulation rate | up to 24 weeks
  The number of follicles that mature and ovulate during a given menstrual or estrous cycle is referred to as ovulation rate or quota.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Mageed M Sarhan, MD, Study Director — Zagazig University
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No